CLINICAL TRIAL: NCT06555003
Title: Comparative Analysis of the Efficacy of Irinotecan-loaded Drug-eluting Beads (DEBIRI) in Combination With Systemic Chemotherapy Versus Chemotherapy Alone in Unresectable Colorectal Cancer Liver Metastases: a Randomized Clinical Trial
Brief Title: DEBIRI Plus Chemotherapy vs. Chemotherapy Alone in Colorectal Cancer Liver Metastases
Acronym: CLEAR-DEBIRI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Jafarian, Professor of General Surgery, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 72101-246-1-1403
Record Dates: First submitted 2024-08-05; First posted 2024-08-15 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Liver Neoplasm; Colorectal Cancer Metastatic
Keywords: irinotecan loaded drug-eluting beads TACE (DEBIRI-TACE); colorectal liver metastases; survival; irinotecan; chemoembolization
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DEBIRI+ Chemotherapy +/- Targeted therapy (Experimental): Patients will receive systemic chemotherapy on day 0 and 14 and DEBIRI on day 7 and 21.
  Interventions: Drug: Drug-Eluting Embolic Bead
- Chemotherapy +/- Targeted therapy (Active Comparator): Patients will receive 4 cycles of systemic chemotherapy.
  Interventions: Drug: Chemotherapy drug

INTERVENTIONS:
Drug: Drug-Eluting Embolic Bead — A minimum of 2 sessions of DEBIRI treatment and 2-4 cycles of systemic chemotherapy are administered (based on tumor size, bilobar or unilobar involvement of the liver, treatment response rate, treatment tolerance, occurrence of side effects, and liver function). Prior to performing DEBIRI, initial angiography is done via the femoral or axillary artery to determine the anatomy of the right and left hepatic arteries as well as the arteries supplying the tumor. Subsequently, a vial of irinotecan (100 mg) eluted with a vial of beads(hepaSphere 25mg) is injected into the blood vessels feeding the tumor. The intervention will be repeated to deliver 200 mg of irinotecan intravascularly to the liver mass. A 14-day interval between the procedures is established to minimize side effects. Targeted therapy administration for each treatment group based on oncologist's decision and will be tailored to the tumor characteristics and the patient's clinical status as explained in control arm.
  Other Names: Irinotecan-loaded drug-eluting beads (DEBIRI) plus systemic chemotherapy +/- targeted therapy
  Arms: DEBIRI+ Chemotherapy +/- Targeted therapy
Drug: Chemotherapy drug — Control group will receive 2-4 cycles of systemic chemotherapy based on functional status of the patient, adverse event rate and treatment tolerance, tumor size and characteristics. Targeted therapy administration for each treatment group in based on oncologist's decision and will be tailored to the tumor characteristics and the patient's clinical status (e.g., administration of Pembrolizumab for patients with high rosatellite instability (MSI-H) or Bevacizumab for tumors harboring KRAS mutations). Due to the targeted nature of these therapies, they can not be administered to all participants of the trial, while It is not ethically justifiable to withhold targeted therapies from patients who are candidates for these treatments based on their tumor characteristics and deprive them of potentially life-extending options.
  Other Names: Systemic chemotherapy +/- targeted therapy
  Arms: Chemotherapy +/- Targeted therapy

SUMMARY:
A total of 116 patients who meet the inclusion criteria and are chemotherapy-naïve for their metastatic disease, will be randomly assigned to either the treatment group (DEBIRI plus systemic chemotherapy) or the control group (systemic chemotherapy alone).

After 4 cycles of chemotherapy and 2 cycles of DEBIRI, patient reassessment to evaluate treatment response, based on RECIST criteria, will be performed using MRI or CT scan within 1-3 months of treatment initiation.

The feasibility of secondary tumor resection, as primary endpoint, will be reassessed at a three-month follow-up multidisciplinary team (MDT) meeting, guided by established clinical guidelines.

DETAILED DESCRIPTION:
Upon acquiring ethical approval, patients with histologically proven, unresectable or borderline resectable liver metastases from colorectal origin who are referred to the hepatobiliary clinic between September 2024 and September 2026 will be enrolled to the study. Informed consent will be obtained for their participation prior to enrollment.

A total of 116 patients who are chemotherapy-naïve for their metastatic disease, will be randomly assigned to either the treatment group or the control group.

With the aim of controlling major confounding factors, Stratified randomization will be performed based on synchronous/metachronous liver metastases and unresectable/borderline resectable status.

Targeted therapy administration for each treatment group in based on oncologist's decision and will be tailored to the tumor's biological characteristics and the patient's clinical status. Ultimately, patients will be categorized into one of the two following treatment groups:

Group 1: DEBIRI+ standard systemic chemotherapy ± Targeted therapy Group 2: Standard systemic chemotherapy ± Targeted therapy The Tumor characteristics, including the number, size, and anatomical location, as well as the presence or absence of extrahepatic metastases, will be assessed based on initial imaging (MRI).

The treatment protocol is defined as the administration of a chemotherapy regimen on days 0 and 14, followed by DEBIRI on days 7 and 21. Each patient of the treatment arm will receive at least two doses of DEBIRI unless treatment-limiting adverse events occur.

After 4 cycles of chemotherapy and 2 cycles of DEBIRI, patient reassessment to evaluate treatment response will be performed using MRI or CT scan within 1-3 months of treatment initiation. All imagings will be reviewed by 2 radiologists who are blinded to clinical information regarding treatment arm. Treatment response will be determined using RECIST criteria.

Conversion to resectability, as primary endpoint, will be evaluated at a three-month follow-up multidisciplinary team (MDT) meeting, guided by established clinical guidelines.

Secondary endpoints of the study will encompass evaluation of treatment tolerability and adverse event rate, alongside analyzing progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* unresectable/borderline resectable colorectal cancer liver metastases, chemotherapy-naïve for metastatic disease, Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less adequate hematologic, hepatic, and renal function ( absolute neutrophil count ≥ 1.5 × 10^9/L, platelet ≥ 75 ×10^9/L, international normalized ratio ≤ 1.3, Total bilirubin ≤ 2.0 mg/dL, aspartate aminotransferase and alanine aminotransferase ≤ 5 × the upper limit of normal (ULN), Albumin ≥ 2.5 g/dL, Creatinine ≤ 2.0 mg/dL)

Exclusion Criteria:

* candidates for curative surgery without the need for neoadjuvant therapy, Liver involvement of ≥ 70%, brain metastases or Peritoneal carcinomatosis, cirrhosis, presence or History of an allergic reaction to any of the study drugs Chronic viral hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Conversion to resectability: The proportion of patients who were initially deemed unresectable but, after undergoing specific intervention (Based on study arm) are reassessed for tumor shrinkage and found to be candidates for surgical resection. | within 3 months after treatment initiation
  The feasibility of secondary tumor resection after receiving treatment, based on follow up imaging and tumor downsizing, will be discussed in multidisciplinary meeting (including surgeons, radiologists and oncologists).

SECONDARY OUTCOMES:
Adverse event rate | Within 1 year of treatment administration
  Unfavorable and unintended signs and symptoms associated with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Jafarian, MD, Principal Investigator — Tehran University of Medical Sciences, Tehran, Iran
Locations (1):
- Imam khomeini hospital complex, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No